CLINICAL TRIAL: NCT01854424
Title: Involvement of Fibrocytes in Repair Processes During Acute Respiratory Distress Syndrome (Validation Study-2)
Brief Title: Validation of the Percentage of Alveolar Fibrocyte as Biomarker During ARDS
Acronym: IFRA2
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: NI11026; AOM 11005 (Other: Assistance publique)
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS); Mechanical Ventilation
Keywords: Fibrocyte; Acute Respiratory Distress Syndrome; Serum Amyloid P; Fibrosis; Mortality
MeSH Terms: conditions — Respiratory Distress Syndrome; Fibrosis | interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients or relatives will be informed of the study. The samples (Bronchoalveolar lavage fluid -BALF-and blood samples) will be obtained in current care and stored in an authorized center of biological resources (CRB Bichat- DC 2009-940)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ARDS: Ventilated patients with ARDS criteria (Berlin criteria) will be recruited in 3 ICU (2 from Bichat Hospital and 1 from Tenon Hospital, Paris) during the first 48 hours of their evolution. The patients will considered in 2 groups during analysis by taking into account their vital status at day-28 of inclusion.
  Interventions: Other: Bronchoalveolar lavage (BAL) before day 2 , between days 5-7 and days 10-14 of evolution.

INTERVENTIONS:
Other: Bronchoalveolar lavage (BAL) before day 2 , between days 5-7 and days 10-14 of evolution. — All the samples will be obtained during current care in the first week of evolution, and the last set of samples (BAL and blood sample between day 10-14) only in patients still under ventilation at this time point.

SUMMARY:
Fibrocyte is a monocyte sub-population involved in fibroproliferation/repair processes and associated with outcome in different diseases. In previous study, we have demonstrated the presence of alveolar fibrocytes during Acute expiratory Distress Syndrome (ARDS) and their association with patient outcome. The purpose of this multicentric observational prospective study is to describe the percentage of alveolar fibrocytes in ICU patients with ARDS (survivors vs. non survivors) and to confirm their association with 28-day mortality.

DETAILED DESCRIPTION:
Background: The acute respiratory distress syndrome (ARDS) remains common (15% of ventilated patients in the ICU), severe (30% of mortality) and have no specific treatment. Impaired epithelial repair with fibroproliferation is observed in non resolutive form of ARDS. Fibrocytes are cells that both express markers of hematopoietic cells (CD34+, CD45+) and fibroblasts (collagen-1). Fibrocytes may be recruited directly from the pool of circulating blood monocytes but also derive from monocytes in situ in absence of serum amyloid P (SAP or pentraxin-2). In murine models of lung injury, it has been shown that fibrocytes were recruited in the lung and contribute to the local fibrogenesis. Our team is the first to have demonstrated during ARDS in human the presence of fibrocytes among the alveolar cells obtained by bronchoalveolar lavage (BAL) (Quesnel et al, Eur Resp J, 2010). In a second single-center work enrolling 122 patients, we have shown that a percentage of alveolar fibrocytes > 6% was associated with an increased risk of death (HR = 6.2 [2.8 to 13.6], p <0.0001). However, this result remains to be confirmed in a second cohort because it was not the main objective of the first study and because of the variable lead time of BAL sampling in this cohort of patients with ARDS (Quesnel et al, CCM, 2012). Furthermore, the correlation of the percentage of blood fibrocytes (Fsg%) with the percentage of alveolar fibrocytes (Fal%) remains unknown and their kinetics remain to be studied during ARDS evolution.

Hypothesis and Objective: We hypothesize that percentage of alveolar fibrocytes is a prognostic marker during ARDS. Our main goal is to confirm in a validation cohort that the % of alveolar fibrocytes measured in BAL fluid during the first 48 hours of ARDS evolution is associated with 28-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* Ventilated patients with ARDS criteria as defined by Berlin criteria during the first 48 hours of evolution.

Exclusion Criteria:

* refusal of patient participation, pregnancy, HIV infection, Respiratory insufficiency, Pulmonary fibrosis, cirrhosis (> Child B score), scleroderma, Alzheimer's disease, Bone marrow transplant, chemotherapy-induced aplasia, immunosuppressive therapy, Corticosteroids (> 200 mg/day of hydrocortisone or equivalent in the two weeks preceding inclusion), End of life patient or IGS2 greater than 90, brain death, therapeutic limitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically Ventilated patients after Sepsis, infectious pneumonia, trauma or postoperative complications.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2013-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07-11 (Actual)

PRIMARY OUTCOMES:
To determine the percentage of alveolar fibrocytes in survivors vs. non survivors during ARDS | alveolar fibrocytes percentage in BALF obtained in the 48 hours following ARDS diagnosis
  Association with 28-day mortality after inclusion

SECONDARY OUTCOMES:
To evaluate kinetics of alveolar and circulating fibrocytes between day-1 and day-14 of ARDS evolution | < day-2, day-3, day 5-7, day 10-14
  number of fibrocytes in BALF and blood samples
To test the prognostic value of the percentage of alveolar fibrocytes during ARDS | < day-2
  Correlation between the percentage of alveolar or blood fibrocytes before day-2 and ventilation time (number of days without invasive ventilation between day 1 and day 28) and length of stay with organ failure (SOFA score evolution between day 1 and 28).
To evaluate the association between the percentage of alveolar fibrocyte and inflammatory and fibroproliferative markers | < day-2, day 5-7, day 10-14
  association between % of alveolar fibrocytes and markers of epithelial injury and fibroproliferation (alveolar and serum IL-8, IL-10, sRAGE, TGF-beta, procollagen III, SAP, CCL18, concentrations) evaluated at day 1, 3, 5-7 and 10-14.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Quesnel, MD, PhD, Principal Investigator — Assistance Publique
Locations (1):
- Hôpital TENON, département d'anesthésie-réanimation, Paris, France